CLINICAL TRIAL: NCT01955499
Title: A Phase I Study of Ibrutinib (PCI-32765) in Combination With Lenalidomide in Relapsed and Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Lenalidomide and Ibrutinib in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01810; NCI-2013-01810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 13022; 9426 (Other: Ohio State University Comprehensive Cancer Center); 9426 (Other: CTEP); K24CA201524 (NIH); P30CA016058 (NIH); U01CA076576 (NIH); U01CA132123 (NIH); UM1CA186644 (NIH); UM1CA186705 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — Specimen Handling; Biopsy; ibrutinib; Lenalidomide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenalidomide, ibrutinib) (Experimental): Patients receive lenalidomide PO on days 1-21 and ibrutinib PO on days 1-28 (days 2-28 of cycle 1). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and CT or PET/CT throughout the study. Patients may undergo bone marrow biopsy and aspiration and MRI as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide and ibrutinib in treating patients with B-cell non-Hodgkin lymphoma that has returned (relapsed) or not responded to treatment (refractory). Lenalidomide helps shrink or slow the growth of non-Hodgkin lymphoma. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving lenalidomide with ibrutinib may work better in treating non-Hodgkin lymphoma than giving either drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of the combination of lenalidomide and ibrutinib in patients with relapsed and refractory B-cell non-Hodgkin's lymphoma (NHL).

II. To define the qualitative and quantitative toxicities of the combination of lenalidomide and ibrutinib.

SECONDARY OBJECTIVES:

I. To describe the overall objective response rate to the combination of lenalidomide and ibrutinib in patients with relapsed or refractory B-cell NHL.

II. To describe the response duration and two-year progression free survival (PFS) in patients with B-cell NHL receiving lenalidomide and ibrutinib.

III. To characterize the pharmacokinetics of the combination of lenalidomide and ibrutinib in patients with relapsed or refractory B-cell NHL.

IV. To identify associations of genetic polymorphisms in drug metabolizing enzymes, transporters or target genes with pharmacokinetics, pharmacodynamics, and clinical outcomes.

V. To monitor the effects of combined therapy with ibrutinib and lenalidomide on B- T-, and natural killer (NK)-cell subsets by flow cytometry and quantitative immunoglobulin levels.

VI. To explore the effects of the combination of ibrutinib and lenalidomide on pharmacodynamic markers including T helper cell, type 1 (TH1) and T helper cell, type 2 (TH2) cytokines, ex vivo NK cell cytotoxicity, serum micro ribonucleic acids (RNAs), plasma metabolites, and levels of Bruton's tyrosine kinase occupancy and other selected kinases.

VII. To explore the relationship between pretreatment pathologic prognostic features and overall objective response.

OUTLINE: This is a dose-escalation study.

Patients receive lenalidomide orally (PO) on days 1-21 and ibrutinib PO on days 1-28 (days 2-28 of cycle 1). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection and CT or PET/CT throughout the study. Patients may undergo bone marrow biopsy and aspiration and MRI as clinically indicated.

After completion of study treatment, patients are followed up for 4 weeks and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell non-Hodgkin's lymphoma (NHL) of any of the following subtypes recognized by the World Health Organization (WHO) classification: diffuse large B-cell lymphoma, mantle cell lymphoma, marginal zone lymphoma, lymphoplasmacytic lymphoma, or follicular lymphoma; patients with evidence of histological transformation to diffuse large B-cell lymphoma from indolent NHL are eligible
* Patients must have received at least one prior therapy; prior autologous stem cell transplant is permitted; patients with diffuse large B-cell lymphoma who have not received high-dose therapy (HDT)/autologous stem cell transplant (ASCT) must be ineligible for HDT/ASCT; prior allogeneic stem cell transplant is not permitted; prior ibrutinib is not permitted
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ibrutinib in combination with lenalidomide in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Patients must have normal organ and marrow function, independent of growth factor or transfusion support; patients should not receive growth factors or transfusions for at least 7 days prior to first dose of study drug, with the exception of pegylated G-CSF (pegfilgrastim) and darbepoeitin which require at least 14 days prior to screening and randomization
* Absolute neutrophil count >= 1,000/mcL in the absence of growth factor administration
* Platelets >= 50,000/mcL in the absence of transfusion support within 7 days prior to determination of eligibility
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilberts disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal unless due to disease
* Creatinine =< 2.0 mg/dL OR creatinine clearance >= 50 mL/min as determined by the Cockcroft-Gault equation or a 24 hour urine collection
* Non-pregnant and non-nursing; due to the known teratogenic potential of lenalidomide and the unknown teratogenic potential of ibrutinib, pregnant or nursing patients may not be enrolled; females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide and for 28 days after the last dose of study drug; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; a FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Patients with human immunodeficiency virus (HIV) infection are eligible provided they meet the following criteria: no evidence of co-infection with hepatitis B or C, cluster of differentiation (CD)4 count >= 400 cells/mm^3, no resistant viral strains, on highly active antiretroviral treatment (HAART) therapy with a viral load < 50 RNA copies/ml, and no history of acquired immunodeficiency syndrome (AIDS)-defining conditions
* Ability to understand and the willingness to sign a written informed consent document
* Curative therapy must have been exhausted or not feasible to administer; patients with diffuse large B-cell lymphoma, germinal center subtype should only enroll on the study if there are no other potentially effective therapeutic options

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; steroids used for disease related symptoms should be stopped within 48 hours of protocol therapy; patients who have had prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor; patients who received monoclonal antibody =< 6 weeks prior to first administration of study treatment
* Patients who are receiving any other investigational agents
* Patients with active central nervous system (CNS) involvement with lymphoma should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to lenalidomide or compounds of similar chemical or biologic composition to lenalidomide including thalidomide
* Patients receiving any medications or substances that are strong inhibitors or strong inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements; currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction, unstable angina or acute coronary syndrome within 6 months prior to randomization
* Recent infections requiring systemic treatment need to have completed therapy > 14 days before the first dose of study drug
* Medications with a risk of causing Torsades de Pointes are not permitted; although concomitant treatment with corrected QT (QTc) prolonging agents is not strictly prohibited, these agents should be avoided whenever possible and an alternative non-QTc prolonging drug should be substituted if possible
* Patients requiring any therapeutic anticoagulation are excluded; patients who have received warfarin or other vitamin K antagonists within 28 days or are taking warfarin or other vitamin K antagonists are not eligible
* Patients who are within 4 weeks of major surgery or within 2 weeks of minor surgery
* Concurrent systemic immunosuppressant therapy other than corticosteroids (e.g. cyclosporine A, tacrolimus, etc) within 28 days of the first dose of study drug
* Vaccinated with live attenuated vaccines within 4 weeks of first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 5), grade =< 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g. von Willebrand's disease) or hemophilia
* Unwilling or unable to participate in all required study evaluations and procedures
* Currently active, clinically significant hepatic impairment (>= moderate hepatic impairment according to the National Cancer Institute (NCI)/Child Pugh classification
* Patients requiring daily corticosteroids at a prednisone equivalent of >= 20 mg daily should not be enrolled; if corticosteroids can be discontinued (or reduced to < 20 mg per day of prednisone or equivalent), the discontinuation or dose reduction should be done at least 7 days prior to first dose
* Unable to swallow capsules, or disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, or symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction
* Serologic status reflecting active hepatitis B or C infection; patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAG), or hepatitis C antibody, must have a negative polymerase chain reaction (PCR) prior to enrollment; (PCR positive patients will be excluded)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days
  Defined as the highest safely tolerated dose where at most one patient experiences dose limiting toxicity (DLT) with the next higher dose having at least 2 patients who experience DLT.
Incidence of toxicity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 criteria | Up to 2 years
  Worst grade toxicities will be recorded for each patient and summarized using frequency tables. Tolerability of the regimen is assessed by summarizing the number of patients who required dose modifications and/or dose delays. In addition, the proportion of patients who go off treatment due to adverse reactions or even those who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial will be counted.

SECONDARY OUTCOMES:
Number of patients responding to treatment | Up to 2 years
  Responses will be summarized with simple descriptive statistics, delineating complete responses from lesser responses and stable disease or progressive disease according to the International Harmonization Project Lymphoma Response Criteria and the Response Criteria for Waldenstrom's Macroglobulinemia.
Degree of response | Up to 2 years
  Responses will be summarized with simple descriptive statistics, delineating complete responses from lesser responses and stable disease or progressive disease according to the International Harmonization Project Lymphoma Response Criteria and the Response Criteria for Waldenstrom's Macroglobulinemia.
Duration of overall response | From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
  Summarized with simple descriptive statistics.
Duration of stable disease | From the start of the treatment until the criteria for progression are met, assessed up to 2 years
  Summarized with simple descriptive statistics.
Progression free survival (PFS) | Duration of time from the start of treatment to the time of measured progression or death, assessed up to 2 years
  Summarized with simple descriptive statistics.

OTHER OUTCOMES:
Pharmacokinetic interactions between lenalidomide and ibrutinib | Baseline and on days 1, 2, and 22 of course 1
  Confidence intervals will be presented as the primary method of analysis.
Single gene polymorphisms, such as those in genes coding for relevant drug metabolizing enzymes, receptors and transporters | Baseline and on day 1 of course 1
  Pharmacogenetic analyses will be conducted to identify single gene polymorphisms and their effects on drug response. Confidence intervals will be presented as the primary method of analysis.
Ki67 staining | Baseline
  Potential relationships with response will be explored using graphical analyses and quantitative summaries. Confidence intervals will be presented as the primary method of analysis.
Change in pharmacodynamic markers including TH1 and TH2 cytokines, ex vivo NK cell cytotoxicity, serum microRNAs, plasma metabolites, and levels of Bruton's tyrosine kinase occupancy and other selected kinases | Baseline, on days 1 and 8 of course 1, and day 1 of courses 2 and 3
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values, and repeated measures analysis of variance will be used to analyze data collected serially over time, recognizing the inherent limitations due to the sample size. Hence, graphical analyses will also be used, including box plots and individual time plots to help identify potential patterns, provide important insights into mechanism, and gather essential preliminary data.
Changes in B- T-, and NK- cell subsets | Baseline and on day 1 of courses 1, 3, 6, and 12
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values, and repeated measures analysis of variance will be used to analyze data collected serially over time, recognizing the inherent limitations due to the sample size. Hence, graphical analyses will also be used, including box plots and individual time plots to help identify potential patterns, provide important insights into mechanism, and gather essential preliminary data.
Changes in quantitative immunoglobulin levels | Baseline and on day 1 of courses 1, 3, 6, and 12
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values, and repeated measures analysis of variance will be used to analyze data collected serially over time, recognizing the inherent limitations due to the sample size. Hence, graphical analyses will also be used, including box plots and individual time plots to help identify potential patterns, provide important insights into mechanism, and gather essential preliminary data.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Christian, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada